CLINICAL TRIAL: NCT05120037
Title: MRI Study of High Definition Transcranial Electrical Stimulation in Chronic Tinnitus (MRI HDtES-T)
Acronym: MRI HDtES-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amber Leaver, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00215708
Record Dates: First submitted 2021-11-12; First posted 2021-11-15 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation (tDCS) uses a mild electrical current to make small (or subtle) changes to how the brain works (or functions).

SUMMARY:
The purpose of this research is to understand how a neurostimulation technique, transcranial electrical stimulation (tES), affects brain function in adults with chronic subjective tinnitus measured with functional magnetic resonance imaging (fMRI). This study targets a specific kind of tES called transcranial direct current stimulation (tDCS), where a mild, constant current is passed between electrodes placed on the scalp.

DETAILED DESCRIPTION:
This is an investigator-initiated MRI study of High Definition (HD) transcranial electrical stimulation (tES) in adults with chronic subjective tinnitus. HDtES is a mild, noninvasive form of brain stimulation using small electrodes to target a small part of the brain/cortex. Primary outcomes are changes in brain function and connectivity measured with MRI before and after a single 20-minute session of HDtES. Secondary outcomes are changes in tinnitus symptoms after 20-minutes of HDtES on 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 75
2. Race/ethnicity: all races and ethnic groups
3. Sex/Gender: all
4. Capacity to provide informed consent
5. Subjective tinnitus symptoms confirmed by patient self report meeting the following criteria:

   1. Present for at least one year prior to start of study
   2. Present (can be heard when consciously attended to) >50% of awake time
   3. Intrudes (is heard even when attempting to ignore/mask) >10% of awake time
6. Has discussed tinnitus symptoms with clinician (i.e., physician, audiologist) to confirm low/no likelihood of physical or neurological origin of tinnitus symptoms (e.g., acoustic neuroma, Meniere's Disease, etc.), confirmed by patient self-report
7. Stable standard or no pharmacological treatment regimen for tinnitus with no change in treatment 6 weeks prior to study start

Exclusion Criteria:

1. Ages below 18 (neurobiology is quite different in children vs. adults)
2. Ages above 75 (cortical excitability changes with age)
3. Tinnitus symptoms with known medial origin, including:

   1. Meniere's disease
   2. Pulsatile tinnitus
   3. Acoustic neuroma
   4. Spontaneous optoacoustic emissions
   5. Any other known medical origin
4. Severe mood disorder (major depression or anxiety)
5. Diagnosis of any medical condition potentially affecting brain function, including:

   1. neuropsychiatric or mental disorders (bipolar, post-traumatic stress disorder, etc.)
   2. severe mood disorders (major depression or anxiety)
   3. psychotic states or disorders
   4. developmental disorders
   5. neurological disorders, including mild cognitive impairment
   6. significant head injury
   7. significant history of alcohol/substance abuse or dependence
   8. active chronic pain condition (>1 year duration)
   9. other major medical conditions (e.g., cancer, stroke).
6. MRI contraindications:

   1. metal or other implants that are not MR-safe
   2. claustrophobia
   3. pregnancy or suspected pregnancy
7. tDCS contraindications*:

   1. skin conditions or injuries on the scalp
   2. hair extensions, wigs, braids, etc. that cannot be removed prior to the study
   3. metal implants or pacemakers (also contraindicated for MRI)
8. Non-English speakers (due to written consent and questionnaires administered)
9. Significant history of alcohol/substance abuse or dependence within last 12 months
10. Neurostimulation or neuromodulation treatment longer than 20 minutes within the past 3 months
11. Current medication use potentially affecting brain function, including decongestants, antihistamines, benzodiazepines or other anticonvulsants, or anti-psychotics.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in brain functional connectivity. | immediate
  Functional MRI will measure changes in brain function during tDCS. Specifically, the investigators will measure change in functional connectivity of prefrontal cortex (% change in Fisher's z).

SECONDARY OUTCOMES:
Changes in tinnitus symptoms | 1 week, 2 weeks, 1 month
  Symptoms of tinnitus will be measured before and after 5 sessions of tDCS using the Tinnitus Functional Index (TFI). Change in TFI scores will be used as a secondary outcome measure. Score range is 0-100, where low scores indicate low symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Translational Imaging at Northwestern University, Chicago, Illinois, United States